CLINICAL TRIAL: NCT03821896
Title: Feasibility, User Experiences, and Preliminary Effectiveness of Conversation Cards for Adolescents, a Patient-centered Communication and Behavior Change Tool: a Pragmatic, Pilot Randomized Controlled Trial
Brief Title: Piloting Conversation Cards for Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Ongoing COVID-19 restrictions and very low (in-person) clinical activity prevented participant recruitment.
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00083903
Record Dates: First submitted 2019-01-18; First posted 2019-01-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-07

CONDITIONS: Adolescent Obesity; Life Style; Health Behavior; Health Communication; Primary Health Care
Keywords: Adolescents; Obesity; Lifestyle; Goals; Communication
MeSH Terms: conditions — Pediatric Obesity; Health Behavior; Obesity; Communication | interventions — Organizational Objectives

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An external party (Women and Children's Health Research Institute, University of Alberta) will run data analysis for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conversation Cards for Adolescents and Goal-Setting (Experimental): Adolescents in the experimental arm will receive the tool 15 minutes prior to their appointment with their primary care provider. They will be instructed to familiarize themselves with the tool and to select the top 3 factors that resonate most with them in their attemps to change their lifestyle habits. They will then proceed to their clinical appointment to set one S.M.A.R.T. goal based on their selections and in collaboration with their primary care provider.
  Interventions: Behavioral: Conversation Cards for Adolescents and Goal-Setting
- Goal-Setting (Active Comparator): Adolescents in the control arm will not complete the tool activity, but will still set a S.M.A.R.T. goal with their primary care provider.
  Interventions: Behavioral: Goal-Setting

INTERVENTIONS:
Behavioral: Conversation Cards for Adolescents and Goal-Setting — The intervention includes using an adolescent-tailored tool (a deck of cards) created by researchers at the University of Alberta and adolescents with obesity seeking weight management care. It contains a list of factors that make it easy or hard for teens to make and maintain healthy lifestyle changes. Its use will be paired with a S.M.A.R.T. goal-setting activity using principles of shared decision-making.
  Arms: Conversation Cards for Adolescents and Goal-Setting
Behavioral: Goal-Setting — Collaborative setting of S.M.A.R.T. goals using principles of shared decision-making.
  Arms: Goal-Setting

SUMMARY:
Providers are not opportunistic enough in addressing lifestyle habits of teens, and can benefit from appropriate tools to support their conversations with families as well as engage all family members in making changes. Since most teens with obesity do not meet minimum lifestyle recommendations, our team developed Conversation Cards for Adolescents (CCAs), a tool to help teens and providers communicate and set lifestyle goals together. In this study, the investigators will (i) observe if and how CCAs fit in a clinical setting for changing teen-provider interactions and teens's lifestyle habits, (ii) ask teens and providers for their thoughts on CCAs and how they are used, and (iii) determine preliminary impact of CCAs on teen behaviors and clinical factors. The investigators will do this with around 50 teens from a primary/secondary care clinic in Edmonton, Alberta. Teens will be randomized to one of two groups - one group will use CCAs in their appointment with their providers to set a goal for change, while the other will also set a goal for change, but without using CCAs. Results from this study will give us insight into how CCAs are best used in a clinical setting and will help us plan a future full-scale study.

DETAILED DESCRIPTION:
Background & Rationale. The high prevalence and adverse health risks of adolescent obesity are well-documented. Most adolescents with and without obesity do not meet minimum lifestyle recommendations for nutrition, physical and sedentary activities, and sleep, and care providers have identified a lack of tools and resources to help them better support families in lifestyle change and weight management. Best practices encourage the use of appropriate tools to augment discussions, in addition to the inclusion and engagement of all relevant stakeholders. Our team conducted a multi-phase project that included adolescents, care providers, and researchers to develop Conversation Cards for Adolescents (CCAs), an adolescent-tailored educational tool aimed at facilitating lifestyle behavior change in adolescents via collaborative goal-setting. This tool comprises a deck of 45 cards. Each card contains an individual statement pertaining to a barrier, enabler, or potential enabler that adolescents encounter in making and maintaining healthy lifestyle changes. These cards are organized across seven categorical suits: nutrition, physical activity, sedentary activity, sleep, mental health, relationships, and clinic factors. This deck is intended to be used by adolescents and providers and may be complementary to an already existing deck of cards (Conversation Cards©) created for parents and providers by our research team in 2012.

Objectives. To (i) assess the feasibility of the study design and procedures in a real-world practice setting, (ii) investigate future trial procedures, (iii) assess user experiences of CCAs, and (iv) determine the preliminary effectiveness of CCAs on changing behavioral and affective-cognitive outcomes for adolescents with obesity.

Method & Methodology. This is a pragmatic, pilot randomized controlled trial. Adolescents will be randomly allocated to one of two groups (CCAs or control) with a 1:1 allocation ratio and using permuted blocks of randomly varied sizes 2 and 4. Participant randomization will be performed in REDCap, based on allocation tables that have been generated and uploaded by the Data Coordinating Centre statistician. REDCap maintains an automated audit trail which includes the assigned study identification number, treatment allocation, and date and time of the transaction. The study coordinator will have access to REDcap onsite to randomize adolescents and will provide corresponding allocations to adolescents. The investigators will follow recommended sample sizes for pilot trials; that is, 25 individuals per trial arm for a total of 50, which gives the main trial a 90% power, 0.2 effect size, and two-sided 5% significance. Assuming a recruitment rate of ~85%, a margin of error for the confidence interval of around 10% was estimated; this recruitment rate is derived from similar randomized controlled trials conducted in a primary care setting surrounding obesity and lifestyle in children and youth. The investigators will adhere to the CONSORT statement for planning, conducting, and reporting pragmatic trials.

Recruitment.

Adolescents - Administrative and clinical (nurse) team members will approach families to gauge interest and obtain verbal consent. If given, the study coordinator on-site (MK) will approach families for more information (e.g., study description, developmental and language eligibility screening) and full consent/assent procedures. On the day of their medical appointment, clinic staff will measure adolescents' height and weight before they see their provider. Providers will be recruited by email or verbal invitation through existing relationships with research team members.

Providers - Researchers leading this study have pre-existing relationships with providers practicing at this center. Researchers will hold several meetings with providers to explain and refine the study and determine their interest in participation. Providers will be given full freedom to accept or decline participation.

The investigators will document dates defining the periods of recruitment and follow-up.

Procedure. Adolescents in the experimental group will be given ~15 minutes before their clinical appointment to review CCAs in a private room at the clinic; they will be instructed to independently select the top 3 statements that most resonate with them and to make a note of these on a provided chart note; these will be documented by the research coordinator on an Excel data file before adolescents enter their appointment and afterwards (in case any changes were made). Adolescents will then proceed to their appointment and collaboratively set one (to facilitate achievement) S.M.A.R.T. (Specific, Measurable, Attainable, Relevant, Time-Based) goal using shared decision-making principles with their provider based on their chosen priorities. Adolescents will receive a hard copy of their specific goal to take home. Adolescents in the control group will not be offered the tool, but will still set a S.M.A.R.T. goal with their provider. The investigators will debrief with each participating provider after their first experimental and first control clinical appointments for feedback and any modifications to intervention procedures.

Outcomes. The study coordinator will create an anonymized detailed Excel data spreadsheet (separate from the Master File) for each participating adolescent to document data. This file will be updated on an ongoing basis. The investigators will collect adolescents' demographic and anthropometric characteristics verbally at baseline and providers' sociodemographics via hard-copy or electronic survey before study commencement. Participants will be instructed to complete baseline outcome measures using an iPad. The investigators will complete 3-week follow-up, where the study coordinator will call adolescents (~15 minutes) for completion of one of the outcome measure assessments and to inquire about study procedures, including ranking the outcome measures used for this study in order of importance (to inform a future full-scale trial). Please refer to the sections below for details regarding outcome measure.

Data Analysis. As per recommendations for pilot studies, our analysis will be mainly of a descriptive nature. Quantitative data will be summarized using quantitative descriptive statistics and central tendencies, or will be compared between groups using independent samples t-tests. Outcomes will be compared based on weight status contingent on anthropometric distributions in our sample. Qualitative data will be audio-recorded, transcribed verbatim using The Comma Police, managed using NVivo 11, and analyzed using content analysis.

Evaluation. The investigators will use the Centers for Disease Control and Prevention Framework for Program Evaluation for a formal evaluation of our intervention. This framework includes engaging stakeholders (e.g., primary users of the evaluation), describing the program (e.g., needs, resources, context, activities), focusing the evaluation design (e.g., purpose, users, questions, methods), gathering credible evidence (e.g., indicators, sources, quality, quantity, logistics), justifying conclusions (e.g., analysis/synthesis, interpretation, recommendations), and ensuring use and shared lessons learned (e.g., design, preparation, feedback, follow-up, dissemination). Steps of this evaluation do not have to occur in a linear sequence; however, earlier steps provide the foundation for subsequent progress. Program evaluations are best completed in a team approach. Our team will include the principal investigator, study coordinator, providers, adolescents, and other researchers in various steps of the evaluation.

IMPLICATIONS. Conducting this research will provide us with lessons learned on how to best use CCAs in a clinical setting. It will inform development of a full scale trial to measure effectiveness of our tool in changing lifestyle behaviors and optimizing care that adolescents receive.

ELIGIBILITY:
Inclusion Criteria:

Adolescents are eligible to participate if they are:

* 13-17 years old
* At a functioning grade level (English literacy and comprehension)
* Interested in setting a lifestyle/behavioural goal related to improving diet, physical activity or sedentary activity, and
* Seeking health services at the Northeast Community Health Centre (NECHC; Edmonton, Alberta, Canada)

All participating providers who deliver care to adolescents at the NECHC are eligible to participate.

Exclusion Criteria:

N/A

Our original eligibility criteria included a BMI ≥85th percentile. After recruiting the first five patients with overweight/obesity from March to August 2019, we decided to remove BMI eligibility criteria given the applicability of our tool's focus on lifestyle and adolescents across the weight spectrum, as well as to enhance recruitment. This decision was made by the research team in conjunction with clinical staff involved in the trial.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Feasibility outcomes for resource, management, and scientific assessments per open-ended questions outlined by Tickle-Degnen's (2013) | Through study completion, an average of 1 year
  The study coordinator will monitor and document study procedures and feasibility based on continuous observation at the site.

SECONDARY OUTCOMES:
Collaborative goal-setting using the Patient Perception of Collaborative Goal-Setting | Baseline
  This questionnaire includes five factors: listen and learn from each other; share ideas; caring relationship; agree on a measurable objective; support for goal achievement. It uses a 5-point scale (worse to better outcome: strongly disagree - disagree - neutral - agree - strongly agree) and has achieved reliability and construct validity. Goal-setting refers to setting one S.M.A.R.T. (specific, measurable, attainable, realistic, timely) goal.
Degree of effort and achievement of treatment goals using researcher-developed questions | 3 weeks
  Questions will use a 0-9 scale (better to worse outcome: 1 - 2 - 3 - 4 - 5 - 6 - 7 - 8 - 9) and will be asked by the study coordinator during the telephone follow-up.
Patient engagement: perspectives on priorities and study design using researcher-developed questions | 3 weeks
  Questions will be open-ended and will be asked by the study coordinator during the telephone follow-up.
Appointment length using a timer on the study-specific iPad | Baseline
  The study coordinator will time the duration of the clinical appointments for both experimental and control groups.
User experience as per the User Experience Questionnaires | Baseline (pre-appt)
  This questionnaire was designed to obtain participants' agreement on contrasting attributes representing gradations between the opposites that may apply to a product. It includes 26 attributes, uses a 7-point scale (better to worse outcome: 1 - 2 - 3 - 4 - 5 - 6 - 7), and has achieved satisfactory reliability and construct validity.
User acceptance as per the Technology Acceptance Model | At study end point, an average of 1 year
  This questionnaire includes 11 items representing perceived usefulness and perceived ease of use of a technology, uses a 7-point scale (better to worse outcome: extremely - quite - slightly - neither - slightly - quite - extremely), and has achieved reliability, internal consistency, and convergent and discriminant validity.
Tool likeability (adolescents) using researcher-developed questions | Baseline
  Questions will be open-ended and closed-ended using a 7-point Likert scale (worse to better outcome: strongly disagree - disagree - somewhat disagree - neutral - somewhat agree - agree - strongly agree)
Tool usefulness (adolescents) using researcher-developed questions | Baseline
  Questions will be open-ended and closed-ended using a 7-point Likert scale (worse to better outcome: strongly disagree - disagree - somewhat disagree - neutral - somewhat agree - agree - strongly agree)
Tool feasibility (adolescents) using researcher-developed questions | Baseline
  Questions will be closed-ended using a 7-point Likert scale (worse to better outcome: strongly disagree - disagree - somewhat disagree - neutral - somewhat agree - agree - strongly agree)
Tool usability (adolescents) using researcher-developed questions | Baseline
  Questions will be closed-ended using a 7-point Likert scale (worse to better outcome: strongly disagree - disagree - somewhat disagree - neutral - somewhat agree - agree - strongly agree)
Tool likeability (PCPs) using researcher-developed questions | At study end point, an average of 1 year
  Questions will be open-ended and closed-ended using a 7-point Likert scale (worse to better outcome: strongly disagree - disagree - somewhat disagree - neutral - somewhat agree - agree - strongly agree)
Tool usefulness (PCPs) using researcher-developed questions | At study end point, an average of 1 year
  Questions will be open-ended and closed-ended using a 7-point Likert scale (worse to better outcome: strongly disagree - disagree - somewhat disagree - neutral - somewhat agree - agree - strongly agree)
Tool feasibility (PCPs) using researcher-developed questions | At study end point, an average of 1 year
  Questions will be closed-ended using a 7-point Likert scale (worse to better outcome: strongly disagree - disagree - somewhat disagree - neutral - somewhat agree - agree - strongly agree)
Tool usability (PCPs) using researcher-developed questions | At study end point, an average of 1 year
  Questions will be closed-ended using a 7-point Likert scale (worse to better outcome: strongly disagree - disagree - somewhat disagree - neutral - somewhat agree - agree - strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Geoff DC Ball, PhD, RD, Principal Investigator — University of Alberta; Maryam Kebbe, PhD, Study Director — University of Alberta
Locations (1):
- Northeast Community Health Centre, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kebbe M, Damanhoury S, Browne N, Dyson MP, McHugh TF, Ball GDC. Barriers to and enablers of healthy lifestyle behaviours in adolescents with obesity: a scoping review and stakeholder consultation. Obes Rev. 2017 Dec;18(12):1439-1453. doi: 10.1111/obr.12602. Epub 2017 Sep 18. PMID 28925065
- [Background] Kebbe M, Perez A, Buchholz A, McHugh TF, Scott SS, Richard C, Mohipp C, Dyson MP, Ball GDC. Barriers and enablers for adopting lifestyle behavior changes in adolescents with obesity: A multi-centre, qualitative study. PLoS One. 2018 Dec 18;13(12):e0209219. doi: 10.1371/journal.pone.0209219. eCollection 2018. PMID 30562377
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Small L, Aplasca A. Child Obesity and Mental Health: A Complex Interaction. Child Adolesc Psychiatr Clin N Am. 2016 Apr;25(2):269-82. doi: 10.1016/j.chc.2015.11.008. Epub 2016 Jan 22. PMID 26980129
- [Background] Skinner AC, Ravanbakht SN, Skelton JA, Perrin EM, Armstrong SC. Prevalence of Obesity and Severe Obesity in US Children, 1999-2016. Pediatrics. 2018 Mar;141(3):e20173459. doi: 10.1542/peds.2017-3459. PMID 29483202
- [Background] Tremblay MS, Feng M, Garriguet D, Ball GDC, Buchholz A, Chanoine JP, Lambert M, Morrison KM. Canadian Pediatric Weight Management Registry (CANPWR): baseline descriptive statistics and comparison to Canadian norms. BMC Obes. 2015 Aug 13;2:29. doi: 10.1186/s40608-015-0060-6. eCollection 2015. PMID 26417450
- [Background] Ball GD, Lenk JM, Barbarich BN, Plotnikoff RC, Fishburne GJ, Mackenzie KA, Willows ND. Overweight children and adolescents referred for weight management: are they meeting lifestyle behaviour recommendations? Appl Physiol Nutr Metab. 2008 Oct;33(5):936-45. doi: 10.1139/H08-088. PMID 18923569
- [Background] Wiegand S, Keller KM, Lob-Corzilius T, Pott W, Reinehr T, Robl M, Stachow R, Tuschy S, Weidanz I, Widhalm K, de Zwaan M, Holl RW. Predicting weight loss and maintenance in overweight/obese pediatric patients. Horm Res Paediatr. 2014;82(6):380-7. doi: 10.1159/000368963. Epub 2014 Dec 20. PMID 25531074
- [Background] He M, Piche L, Clarson CL, Callaghan C, Harris SB. Childhood overweight and obesity management: A national perspective of primary health care providers' views, practices, perceived barriers and needs. Paediatr Child Health. 2010 Sep;15(7):419-26. doi: 10.1093/pch/15.7.419. PMID 21886445
- [Background] McPherson AC, Hamilton J, Kingsnorth S, Knibbe TJ, Peters M, Swift JA, Krog K, Chen L, Steinberg A, Ball GD. Communicating with children and families about obesity and weight-related topics: a scoping review of best practices. Obes Rev. 2017 Feb;18(2):164-182. doi: 10.1111/obr.12485. Epub 2016 Nov 26. PMID 27888564
- [Background] Ball GD, Farnesi BC, Newton AS, Holt NL, Geller J, Sharma AM, Johnson ST, Matteson CL, Finegood DT. Join the conversation! The development and preliminary application of conversation cards in pediatric weight management. J Nutr Educ Behav. 2013 Sep-Oct;45(5):476-8. doi: 10.1016/j.jneb.2013.02.002. Epub 2013 Apr 19. No abstract available. PMID 23602164
- [Background] Arnold DM, Burns KE, Adhikari NK, Kho ME, Meade MO, Cook DJ; McMaster Critical Care Interest Group. The design and interpretation of pilot trials in clinical research in critical care. Crit Care Med. 2009 Jan;37(1 Suppl):S69-74. doi: 10.1097/CCM.0b013e3181920e33. PMID 19104228
- [Background] Schwartz D, Lellouch J. Explanatory and pragmatic attitudes in therapeutical trials. J Clin Epidemiol. 2009 May;62(5):499-505. doi: 10.1016/j.jclinepi.2009.01.012. PMID 19348976
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Thorpe KE, Zwarenstein M, Oxman AD, Treweek S, Furberg CD, Altman DG, Tunis S, Bergel E, Harvey I, Magid DJ, Chalkidou K. A pragmatic-explanatory continuum indicator summary (PRECIS): a tool to help trial designers. J Clin Epidemiol. 2009 May;62(5):464-75. doi: 10.1016/j.jclinepi.2008.12.011. PMID 19348971
- [Background] Treweek S, Lockhart P, Pitkethly M, Cook JA, Kjeldstrom M, Johansen M, Taskila TK, Sullivan FM, Wilson S, Jackson C, Jones R, Mitchell ED. Methods to improve recruitment to randomised controlled trials: Cochrane systematic review and meta-analysis. BMJ Open. 2013 Feb 7;3(2):e002360. doi: 10.1136/bmjopen-2012-002360. Print 2013. PMID 23396504
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Derived] Kebbe M, Farmer A, Dyson MP, Scott SD, McHugh TLF, Lappa S, Rajani H, Ladha T, Islam B, Jacoby L, Nasir F, Talwar K, Wincott JL, Zhang M, Ball GDC. Feasibility, user experiences, and preliminary effect of Conversation Cards for Adolescents(c) on collaborative goal-setting and behavior change: protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2019 Dec 18;5:149. doi: 10.1186/s40814-019-0533-3. eCollection 2019. PMID 31890261